CLINICAL TRIAL: NCT06578000
Title: Efficacy of Iontophoresis in Treating Lateral Epicondylitis Patients a Randomised Controlled Trial
Brief Title: Efficacy of Iontophoresis in Treating Lateral Epicondylitis Patients
Acronym: Iontophoresis
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: NOUR ALI ABO EL ELAA FRAGHLY (Other)
Collaborators: Cairo University (Other)
Responsible Party: Sponsor-Investigator, NOUR ALI ABO EL ELAA FRAGHLY, Lecturer assistant, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: P.T.REC/012/004798
Record Dates: First submitted 2024-08-21; First posted 2024-08-29 (Actual); Last update posted 2024-08-29 (Actual); Status verified 2024-08

CONDITIONS: Lateral Epicondylitis
Keywords: iontophoresis
MeSH Terms: conditions — Tennis Elbow | interventions — Magnesium Sulfate

STUDY DESIGN:
Intervention Model Description: Patients will be assigned randomly into 2 groups:
  Group (A): Iontophoresis therapy (MgO4 will be applied to the active positive electrode and the treatment will be repeated twice a week for four weeks) + traditional therapy (Splint + Stretch + strength).
  Group (B): conventional therapy (Splint + Stretch + strength) twice a week for six weeks
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- group 1 ( Iontophoresis therapy (MgO4 will be applied to the active positive electrode)) (Active Comparator): Iontophoresis therapy (MgO4 will be applied to the active positive electrode and the treatment will be repeated twice a week for four weeks) + conventional therapy (Splint + Stretch + strength).
  Interventions: Drug: Magnesium sulfate; Other: conventional therapy
- Control Group (2): conventional physical therapy treatment (Sham Comparator): conventional therapy (Splint + Stretch + strength) twice a week for six weeks
  Interventions: Other: conventional therapy

INTERVENTIONS:
Drug: Magnesium sulfate — Iontophoresis therapy (MgO4 will be applied to the active positive electrode and the treatment will be repeated twice a week for four weeks) + conventional therapy (Splint + Stretch + strength).
  Arms: group 1 ( Iontophoresis therapy (MgO4 will be applied to the active positive electrode))
Other: conventional therapy — conventional therapy (Splint + Stretch + strength) twice a week for six weeks

SUMMARY:
This study is conducted To evaluate the effect of magnesium sulfate on pain intensity, muscle power, hand grip and function ability in patients with lateral epicondylitis.

DETAILED DESCRIPTION:
This study is conducted To evaluate the effect of magnesium sulfate on pain intensity, muscle power, hand grip and function ability in patients with lateral epicondylitis.

BACKGROUND:

Lateral epicondylitis (LE) (tennis elbow) is a tendinopathy of the forearm extensor muscles, often caused by overuse or repetitive use (mostly of the extensor carpi radialis brevis), forced extension or direct trauma in the epicondyle . LE has an approximate rate of 40% and a prevalence of 1-3% of the general population . It mostly affects people 40 years and older. Some studies indicate that men and women are equally affected; others report a higher percentage of affected women .

HYPOTHESES

It will be hypothesized that:

There will be no statistically significant effect of magnesium sulfate on pain intensity, muscle power, hand grip and function ability in patients with lateral epicondylitis.

Definition of terms Lateral epicondylitis: pain and tenderness over the lateral epicondyle of the humerus, and pain on resisted dorsiflexion of the wrist, middle finger, or both .

Iontophoresis: is a technique used to enhance transdermal penetration of substances through the application of electric current .

RESEARCH QUESTION:

This study will be conducted to answer the following question:

What is the effect of magnesium sulfate on pain intensity, muscle power, hand grip and function ability in patients with lateral epicondylitis?

ELIGIBILITY:
Inclusion Criteria:

* • Their age will be ranged between 20-50 years with both gender

  * Pain on the lateral side of the elbow for at least 4 weeks
  * Tenderness over the lateral epicondyle
  * At least two positive provocative tests: Mill test and Thomson test

Exclusion Criteria:

* • History of injection, surgery, physical therapy in the elbow area in the last 3 months

  * Previous elbow surgery
  * History of radius/ulna fracture
  * History of cervical and shoulder problems
  * Having bilateral symptoms
  * Concomitant medial epicondylitis
  * Malignancy
  * Pregnancy
  * Systemic rheumatologic disease or systemic infection
  * Inserted cardiac pacemaker
  * Presence of coagulation disorders
  * Cognitive dysfunction

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2024-11-30 (Estimated); Study Completion 2025-03-02 (Estimated)

PRIMARY OUTCOMES:
to investigate the effect of magnesium sulfate on pain intensity | 6 weeks
  . Visual analogue scale will be used to assess the pain intensity level. Pain intensity Level will be measured using the VAS that consists of a 10-cm straight line with endpoints defining pain intensity.All patients will be asked to mark their pain level that corresponds to their pain intensity on the line between "0", representing "no pain", and "10", representing "the worst pain imaginable". The distance between "0" and the mark made by the patients was measured. Difference in pain intensity will be recorded at rest, at night, and during activity (repeated elbow movement) at baseline and after treatment
investigate the effect of magnesium sulfate on muscle power in patients with lateral epicondylitis. | 6 weeks
  Cyriax Resisted Muscle Test: In this test, the patients will be seated and positioned with their upper extremities relaxed. The test will include elbow extension, third finger extension, pronation, and supination. All tests were conducted in a standardized manner using maximal isometric resistance and allowing no movement at either joint. Based on manual muscle testing principles, the examiner will hold the contraction for approximately 3 s to allow the patients time to build to maximum tension. The examiner will stabilize the patients' elbows with one hand and applied resistance with other hand. The patients will be instructed to report the onset of or an increase in pain. The results of the resisted tests will be recorded as "strong and painless", "strong and painful", "weak and painful", and "weak and painless". The Cyriax Resisted Muscle Test was conducted at baseline and after treatment
investigate the effect of magnesium sulfate on hand grip in patients with lateral epicondylitis. | 6 weeks
  Maximum grip strength: by using hand dynamometer the patients will be seated on an armless chair with 90° flexion of hip and knee, their shoulders with 0° abduction and in the neutral position, their elbow at 90° flexion and their forearm in the neutral position, and their wrist in semi pronation with an upright thumb to provide a stronger grip. The protocol will consist of three maximal isometric contractions without pain for 5 s with a rest period of at least 60 s. The patients will perform three trials of grip strength using their involved and non-involved hands while maintaining 90° elbow flexion and neutral forearm position. The patients followed a verbal command of "slowly push, push, push, push, and relax" for each isometric contraction to ensure that the contractions lasted for approximately 5 s. The patients will be also asked to squeeze the dynamometer as hard as possible without the sensation of pain. The mean strength of three measurements will be recorded in kilograms
investigate the effect of magnesium sulfate on function ability in patients with lateral epicondylitis. | 6 weeks
  The elbow functionality will be determined using the Patient-Rated Tennis Elbow Evaluation Scale (PRTEE) appendix II. The PRTEE is a 15-item questionnaire designed to measure forearm pain and disability in patients with lateral epicondylitis. The patients must rate their levels of pain and disability from 0 to 10. There are two subscales: the pain subscale (0 = no pain, 10 = worst pain imaginable) and the function subscale (0 = no difficulty, 10 = unable to do)

SECONDARY OUTCOMES:
Elbow range of motion | 6 weeks
  Joint range of motion evaluation: With the wrist in neutral position, the angle achieved during maximum wrist extension was assessed using the Clinometer (Plaincode Software Solution, Stephanskirchen, Germany) which is a smartphone application.
  The forearm placed on the chair armrest, with 90 degrees of elbow flexion, the angle between the radius and the second metacarpal was measured by the radial styloid axis of the forearm in pronation. The interrater reliability for angular measurements was 0.76-0.95 (Lim and Shin, 2016).

CONTACTS AND LOCATIONS:
Overall Officials: Neveen Abd El latif Abdel Raoof, professor, Study Director — Professor of Physical Therapy department for Basic sciences
Locations (1):
- Faculty of Physical Therapy, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided